CLINICAL TRIAL: NCT02600000
Title: Effectiveness of Inspiratory Muscle Training Associated With a Cardiac Rehabilitation Program in Sympathetic Activity and Functional Capacity in Patients With Heart Failure: a Randomized Clinical Trial
Brief Title: Inspiratory Muscle Training Effectiveness in Sympathetic Activity and Functional Capacity in Patients With Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Jéssica Costa Leite, Master's Degree student, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 38572614.1.3001.5192
Record Dates: First submitted 2015-11-04; First posted 2015-11-09 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Exercise Test

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sympathetic myocardial activity after IMT (Experimental): Evaluate the effectiveness of Muscle Training Inspiratory associated with a cardiac rehabilitation program in the modulation of sympathetic myocardial activity of patients with HF
  Interventions: Radiation: Myocardial scintigraphy
- Maximal functional capacity after IMT (Experimental): Evaluate the effectiveness of Muscle Training Inspiratory associated with a cardiac rehabilitation program in the maximal functional capacity of patients with HF
  Interventions: Device: Cardiopulmonary test
- submaximal functional capacity after IMT (Experimental): Evaluate the effectiveness of Muscle Training Inspiratory associated with a cardiac rehabilitation program in the submaximal functional capacity of patients with HF
  Interventions: Device: AVD-Glittre Test
- Thickness and mobility of the diaphragm after IMT (Experimental): Assess the impact of Inspiratory Muscle Training in combination with a cardiac rehabilitation program on the thickness and mobility of the diaphragm in patients with heart failure.
  Interventions: Device: Diaphragm ultrasound

INTERVENTIONS:
Radiation: Myocardial scintigraphy — Myocardial scintigraphy with Iodo123-Metaiodobenzylguanidine (MIBG) to assess the Sympathetic myocardial activity
  Arms: Sympathetic myocardial activity after IMT
Device: Cardiopulmonary test — Assessment of maximal functional capacity
  Arms: Maximal functional capacity after IMT
Device: AVD-Glittre Test — Evaluation of submaximal functional capacity after inspiratory muscle training.
  Arms: submaximal functional capacity after IMT
Device: Diaphragm ultrasound — Evaluation of thickness and diaphragmatic mobility
  Arms: Thickness and mobility of the diaphragm after IMT

SUMMARY:
Heart failure (HF) is configured major problem for public health in the country. Affected individuals may experience fatigue, dyspnea, respiratory muscle weakness, overstimulation of the sympathetic myocardial activity, among others. In relation to the treatment of patients with heart failure with symptoms mentioned above a great alternative is the implantation of cardiac rehabilitation programs, these programs can also be associated with other muscle training measures, among these there is inspiratory muscle training (IMT), as the weakness of these muscles is rather found in this population and this directly related to signs and symptoms. OBJECTIVE: To evaluate the efficacy of inspiratory muscle training associated with a cardiac rehabilitation program in the modulation of sympathetic myocardial activity and maximal and submaximal functional capacity of patients with HF between 21-60 years. METHODOLOGY: This is a clinical trial, controlled, randomized, double-blind being developed in partnership with the Department of Physical Therapy, Federal University of Pernambuco (UFPE) and the Hospital das Clinicas (HC) of Pernambuco, whose patients will be accrued on the Recife's main referral centers in caring for patients with heart failure. Patients will undergo the evaluation of pulmonary function and respiratory muscle strength (spirometry and digital Manovacuometry) as well as on the functional capacity (Ergospirometry), cardiac innervation (myocardial scintigraphy), mobility and diaphragm thickness (ultrasound) and quality of life. After the evaluation will be randomly allocated into two groups: The control group will perform cardiac rehabilitation associated with the Sham of IMT, and the experimental group cardiac rehabilitation associated with the IMT at 30% of maximal inspiratory pressure. The intervention will last three months for both groups and after this phase patients will be submitted again to the assessment tools. EXPECTED RESULTS: To clarify the association between physical exercise associated with specific respiratory training in modulating the autonomic nervous system of patients with HF and what the relationship with reflected cardiorespiratory fitness in maximal and submaximal functional capacity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Heart Failure;
* Lower left ventricular ejection fraction 45% (LVEF <45%) assessed by simple and recent echocardiogram;
* Functional Class II and III by the New York Heart Association (NYHA)
* Clinically stable;
* Ex-smokers over five years;
* Maximal inspiratory pressure (MIP) <70% of predicted;
* Forced expiratory volume/Forced vital capacity (FEV1 / FVC) > 70% of predicted;

Exclusion Criteria:

* Unstable angina;
* Myocardial infarction and heart surgery up to three months before the survey;
* Chronic respiratory diseases;
* Hemodynamic instability;
* Trauma recent face, nausea and vomiting.
* Orthopedic and neurological diseases that may preclude the achievement of the cardiopulmonary test and Cardiac Rehabilitation exercises;
* Psychological and / or cognitive impairments that restrict them to respond to questionnaires;

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-02; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Adrenergic tone of the heart muscle | Change from Baseline and Three months after
  Measured by the integrity and activity of the sympathetic nervous pre synaptic terminals.
Change from Functional capacity | Change from Baseline and Three months after
  Measured by cardiopulmonary exercise testing

SECONDARY OUTCOMES:
Change from Submaximal functional capacity | Change from Baseline and Three months after
  Measured by Glittre Test
Mobility of the diaphragm | Change from Baseline and Three months after
  Reviewed from the ultrasound
Diaphragm thickness | Change from Baseline and Three months after
  Reviewed from the ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Physiology laboratory and cardiopulmonary physiotherapy, Recife, Pernambuco, Brazil

REFERENCES:
- [Derived] Leite JC, Brandao DC, Brandao SCS, Fuzari HKB, Vidal TM, Frutuoso J, Remigio MI, de Araujo BTS, Campos SL, Dornelas de Andrade A. Effectiveness of inspiratory muscle training associated with a cardiac rehabilitation program on sympathetic activity and functional capacity in patients with heart failure: a study protocol for a randomized controlled trial. Trials. 2020 Jun 12;21(1):519. doi: 10.1186/s13063-020-04363-6. PMID 32532283